CLINICAL TRIAL: NCT06264180
Title: Randomized, Ph3 Clinical Study Comparing Vusolimogene Oderparepvec in Combination With Nivolumab Vs Treatment of Physician's Choice in Patients With Advanced Melanoma That Progressed on Anti-PD-1 and Anti-CTLA-4 Containing Treatment [IGNYTE-3]
Brief Title: VO and Nivolumab vs Physician's Choice in Advanced Melanoma That Progressed on Anti-PD-1 & Anti-CTLA-4 Drugs [IGNYTE-3]
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP1-104
Record Dates: First submitted 2024-01-29; First posted 2024-02-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Nivolumab; relatlimab; Opdualag; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VO + nivolumab (Experimental)
  Interventions: Biological: Vusolimogene Oderparepvec; Biological: Nivolumab
- Physicians Choice (Active Comparator): Choosing from 1 of the following (to be consistent with approved label and/or applicable local clinical guidelines):
  * Nivolumab + relatlimab (as Opdualag)
  * Anti-PD-1 monotherapy (nivolumab or pembrolizumab)
  * Single-agent chemotherapy (dacarbazine, temozolomide, or paclitaxel/albumin-bound paclitaxel)
  Interventions: Biological: Nivolumab; Biological: Nivolumab + Relatlimab; Biological: Pembrolizumab; Drug: Single-agent chemotherapy

INTERVENTIONS:
Biological: Vusolimogene Oderparepvec — Genetically modified Herpes Simplex Type 1 Virus.
  Other Names: VO; RP1
  Arms: VO + nivolumab
Biological: Nivolumab — Anti-PD-1 Monoclonal Antibody
  Other Names: Opdivo
Biological: Nivolumab + Relatlimab — Nivolumab: Anti-PD-1 Monoclonal antibody. Relatlimab: A lymphocyte activation gene-3 (LAG-3) blocking antibody.
  Other Names: Opdualag
  Arms: Physicians Choice
Biological: Pembrolizumab — A programmed death receptor-1 (PD-1)-blocking antibody indicated.
  Other Names: Keytruda
  Arms: Physicians Choice
Drug: Single-agent chemotherapy — Dacarbazine, temozolomide, or paclitaxel/albumin-bound paclitaxel.
  Arms: Physicians Choice

SUMMARY:
This is a randomized, controlled, multicenter, open-label Phase 3 clinical study comparing VO in combination with nivolumab versus Physician's Choice treatment for patients with unresectable Stage IIIb-IV cutaneous melanoma whose disease progressed on an anti PD-1 and an anti-CTLA-4 containing regimen (administered either as a combination regimen or in sequence) or who are not candidates for treatment with an anti-CTLA-4 therapy.

ELIGIBILITY:
Key Inclusion Criteria:

I 1. Male or female who is 12 years of age or older at the time of signed informed consent.

I 2. Patients with histologically or cytologically confirmed unresectable or metastatic Stage IIIb through IV/M1a through M1d cutaneous melanoma, as per AJCC staging system, 8th edition).

I 3. Confirmed disease progression (PD) on an anti-PD-1 antibody treatment and an anti-CTLA-4 antibody treatment, administered as either a combination regimen (eg, nivolumab + ipilimumab) or in sequence.

1. Treatment with prior anti-PD-1 therapy must have continued for a minimum of 8 weeks (note: treatment with prior pembrolizumab therapy when administered every 6 weeks must have continued for a minimum of 12 weeks [ie, 2 treatment cycles]). Any number of doses of prior anti-CTLA-4 therapy may have been administered in combination with an anti-PD-1. The anti-PD-1-containing therapy must be the immediate prior line of treatment before randomization (for patients with BRAF mutation, see I 4).
2. Patients who in the physician's judgement are not candidates for treatment with an anti-CTLA-4 antibody (eg, due to documented clinically significant comorbidities or history of immune-related adverse events) are eligible for the study if they have confirmed PD on an anti-PD-1 antibody (including unresectable disease relapse during adjuvant therapy or < 6 months from completion of adjuvant therapy).
3. Disease progression must have been confirmed and documented using clinical or radiological assessment by 2 assessments at least 4 weeks apart while being treated with an anti-PD-1 antibody and an anti-CTLA-4 antibody. Radiological confirmation of PD can occur during the Screening period for this study. Treatment with prior anti-PD-1 therapy must have continued from the time of initial tumor progression until confirmation of PD (ie, such that no doses of anti-PD-1 therapy were missed).

Note: If radiographic progression at the initial scan where PD was documented is accompanied by clear clinical progression, defined as a decline in performance status directly attributed to disease or increased disease-related symptoms, anti-PD-1 therapy does not need to continue. For patients with documented PD while on adjuvant therapy with an anti-PD-1 therapy, a confirmatory biopsy can be used in place of a confirmatory scan.

I 4. Has documented BRAF V600 mutation status or must consent to BRAF V600 mutation testing per local institutional standards during the Screening period. Patients with BRAF mutation should have received prior BRAF-directed therapy (with or without a MEK inhibitor) prior to randomization, unless deemed not clinically indicated at Investigator's discretion due to concurrent medical condition or prior toxicity.

Note: Prior exposure to BRAF-directed therapy (with or without a MEK inhibitor) includes treatment in the adjuvant setting. One line of BRAF-directed therapy (with or without a MEK inhibitor) can be the most recent systemic treatment administered before randomization.

I 5. Has least 1 measurable tumor of ≥ 1 cm in longest diameter (or shortest diameter for lymph nodes) and injectable lesion(s) of at least 1 cm in longest diameter.

I 6. Has adequate hematologic function, including:

1. White blood cell (WBC) count ≥ 2.0 × 109/L
2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
3. Platelet count ≥ 75 × 109/L
4. Hemoglobin ≥ 8 g/dL (without packed red blood cell [RBC] transfusion within 2 weeks of dosing)

I 7. Has adequate hepatic function, including:

1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN; < 2.0 × ULN for patients with known Gilbert syndrome or liver metastases)
2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 × ULN (or ≤ 5.0 × ULN, if liver metastases are present)
3. Alkaline phosphatase (ALP) ≤ 2.5 × ULN (or ≤ 5.0 × ULN, if liver or bone metastases are present) I 8. Has adequate renal function, defined as serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 3 0 mL/minute/1.73 m2 (measured using Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).

I 9. Prothrombin time (PT) ≤ 1.5 × ULN (or international normalization ratio [INR] ≤ 1.3) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Note: Patients who are on chronic anticoagulant therapy may be randomized if the target INR is ≤ 2.5. For patients requiring deep injection of VO, the INR must be <1.5 at the time of injection.

I 10. ECOG performance status (PS) 0 to 1 for patients 18 and older or a Lansky PS ≥ 80 for patients 12 to 17 years of age.

I 11. Life expectancy of at least 3 months. I 12. Female and male patients of reproductive potential must agree to avoid becoming pregnant or impregnating a partner and adhere to highly effective contraception requirements during the treatment period and for at least 6 months after the last dose of any study treatment.

I 13. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units or β hCG within 7 days before the first dose of study treatment.

I 14. Capable of giving signed informed consent which includes willingness to comply with the requirements and restrictions listed in the informed consent form (ICF)

Key Exclusion Criteria:

E 1. Primary mucosal or uveal melanoma. E 2. More than 2 lines of systemic therapy for advanced melanoma. Note: One additional line of anti-PD-1 therapy in the adjuvant or neoadjuvant setting is allowed if the patient was free of treatment and of PD for at least 6 months and subsequently had confirmed PD on an anti-PD-1 and an anti-CTLA-4 antibody therapy administered in the advanced setting.

E 3. Known acute or chronic hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known acute or chronic hepatitis C virus (defined as HCV RNA [qualitative] is detected).

Note: Patients who have been effectively treated are eligible for randomization. Patients must be negative for HBsAg and HCV RNA.

E 4. Known human immunodeficiency virus (HIV) infection. Note: Testing for HIV is not required unless mandated by local health authority or clinically indicated.

E 5. Active significant herpetic infections or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis) or requires intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).

Note: Patients with sporadic cold sores may be randomized if no active cold sores are present at the time of first dose of study treatment.

E 6. Had systemic infection requiring IV antibiotics or other serious active infection requiring antimicrobial, antiviral, or antifungal treatment within 14 days prior to the first dose.

E 7. Evidence of spinal cord compression or at high risk of spinal cord compression.

E 8. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis at time of screening. Patients with known central nervous system metastases are eligible if they have received standard-of-care therapy for central nervous system disease (such as stereotactic radiosurgery or radical surgical resection followed by radiotherapy) and have evidence of disease stability on 2 subsequent scans performed at least at a 4-week interval.

E 9. Serum lactate dehydrogenase (LDH) > 2 × ULN. E 10. Major surgery ≤ 2 weeks prior to starting study treatment. Note: Patients must have recovered adequately from all acute complications of all previous procedures prior to randomization.

E 11. Prior malignancy active within the previous 3 years, except for locally curable cancers that have apparently been cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ (without invasive component) of the prostate, cervix, or breast.

E 12. History of significant cardiac disease including myocarditis or congestive heart failure (defined as New York Heart Association Functional Classification III or IV), or unstable angina, serious uncontrolled cardiac arrhythmia, cerebral vascular accident, or myocardial infarction within 6 months from first dose of VO.

E 13. History of life-threatening toxicity related to prior immune therapy except those that are unlikely to recur with standard countermeasures (eg, hormone replacement after adrenal crisis).

E 14. History or evidence of psychiatric, substance abuse (including IV substance abuse), or any other clinically significant disorder, condition, or disease (with the exception of those described above) that, in the opinion of the Investigator or the Medical Monitor, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.

E 15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

E 16. Active, known, or suspected autoimmune disease requiring systemic treatment.

E 17. History of (noninfectious) pneumonitis that required steroids or has current pneumonitis.

E 18. Prior oncolytic virus therapy or other therapy given by intratumoral administration.

E 19. Requires chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).

E 20. Has received a live vaccine within 28 days prior to the first dose of study treatment.

E 21. Systemic anticancer therapies within 5 half-lives or 4 weeks of the first dose, whichever is shorter.

E 22. Is currently participating in or has participated in a study of an investigational agent within 4 weeks prior to the first dose of study treatment.

E 23. Has received prior radiotherapy within 2 weeks of start of study treatment or has not recovered from radiotherapy.

E 24. Conditions requiring treatment with immunosuppressive doses (> 10 mg per day of prednisone or equivalent) of systemic corticosteroids other than for corticosteroid replacement therapy 14 days before randomization.

Note: Patients who require a brief course (≤ 7 days) or corticosteroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. Physiologic replacement doses of systemic corticosteroids are permitted, only if the dose does not exceed 10 mg/day prednisone equivalent.

E 25. History of allergy or sensitivity to study drug components (VO, nivolumab, pembrolizumab, or relatlimab) or to cisplatin or carboplatin or paclitaxel (dependent on cohort) or prior monoclonal antibody treatment.

E 26. Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to treatment.

E 27. Is a person who is deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2034-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Assessed up to January 2029, approximately 55 months
  Time from the date of randomization to death due to any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Assessed up to January 2029, approximately 55 months
  The time from the date of randomization to the earliest date of the objective documentation of progressive disease (PD) per RECIST v1.1 or death due to any cause.
Objective Response Rate (ORR) | Assessed up to January 2029, approximately 55 months
  The proportion of randomized patients with best overall response of complete response (CR) or partial response (PR) using the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gullo, MD, Study Director — Replimune Inc.
Locations (69):
- United States (49):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - UC Irvine Health, Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Sutter Medical Group, Sacramento, California
  - San Francisco Oncology Associates, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville Brown Cancer Center, Louisville, Kentucky
  - Henry Ford Cancer - Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth Hitchcock Cancer Center, Lebanon, New Hampshire
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health, R.J. Zuckerberg Cancer Center, Lake Success, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University- Martha Morehouse Tower, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - West Cancer Center and Research Institute, Germantown, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Texas Oncology, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Intermountain Health, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - St. George Regional Hospital, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University, Morgantown, West Virginia
- France (4):
  - Hopital de La Timone, Marseille
  - Hôpital Saint Louis - AP-HP, Paris
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Klinik, Erfurt
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Medical Center, Hamburg
  - Universitätsklinikum Hospital Heidelberg, Heidelberg
  - Universitatsklinikum Mainz Hautklinik und Poliklinik, Mainz
  - Universitätsklinikum of Tübingen, Tübingen
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
- The Royal Marsden NHS Foundation Trust, London, United Kingdom